CLINICAL TRIAL: NCT01617057
Title: Therapeutic Efficacy of Tiludronic Acid on Inner Ear Involvement in Advanced Otosclerosis
Acronym: OTOPHOS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P081235
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Otosclerosis
Keywords: otosclerosis; inner ear; tiludronic acid
MeSH Terms: conditions — Otosclerosis | interventions — tiludronic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skelid (Experimental): tiludronic acid
  Interventions: Drug: tiludronic acid
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tiludronic acid — 400 mg / day for 3 months
  Arms: Skelid
Drug: Placebo — 400 mg / day for 3 month
  Arms: Control

SUMMARY:
The aim of this study is to assess the efficacy of a biphosphonate (tiludronic acid, Skelid®, Sanofi-Aventis) in the treatment of inner ear involvement in advanced otosclerosis

DETAILED DESCRIPTION:
Otosclerosis is a bone dystrophy localized to middle and inner ears with unknown etiology. It principally concerns adult patients between 30 and 50 years of age. Women present with this disease 2 times more frequently than men. Family cases are observed in 50% with a dominant autosomal transmission and low penetrance (40%). In its early stages, the disease is mainly located at the stapediovestibular joint leading to its ankylosis and a conductive hearing loss. In its advanced stages, the lesions extend around the cochlea and vestibule, induce a sensorineural hearing loss which can progress to severe and profound deafness, and prolonged balance disorders. On CT-scan, disease foci show a demineralization. Their density is inversely correlated to the hearing loss. In early stage, hearing function is currently rehabilitated by conventional hearing aids or surgery. In advanced forms, cochlear involvement is not accessible to surgery, and rehabilitation is insured by he hearing aids or cochlear implants. Vestibular dysfunction is dealt with by physiotherapy or symptomatic treatment. Drugs with anabolic activity in bone, such as sodium fluoride and etidronate (first generation bisphosphonate, Didronel ®), appear to reduce the hearing loss and to increase the radiological density of disease foci. However, their efficacy is low and poorly documented. Their effect on vestibular function is unknown.

Moreover, ototoxicity has been reported for etidronate. New biphosphonates such as tiludronic acid (Skelid ®) have a significantly more potent inhibition of bone resorption and do not have an ototoxic effect. They have been used for the treatment or the prevention of postmenopausal osteoporosis and in Paget's disease with mild to moderate adverse effects in the majority of cases.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* French citizen
* Signed consent for participation
* No dental infection
* No programmed dental surgery during the treatment
* Effective contraception for women of childbearing potential
* Patient with advanced otosclerosis defined by:
* Slowly progressive uni or bilateral hearing loss
* No past medical history of chronic otitis media
* No past medical history of other causes of cochlear damage (significant surgical trauma with a 30 dB deterioration of bone conduction at 4000 Hz in postoperative period, sound trauma, barotrauma, ototoxic drugs)
* Normal tympanic membranes
* A conductive or mixed hearing loss
* A moderate to severe hearing loss on at least one ear (average of thresholds at 500, 1000, 2000 and 4000 Hz) on air conduction between 30 and 90 dB.
* Normal tympanometry or with a decreased peak
* Absent ipsilateral stapedial reflex
* As possible, intraoperative confirmation of stapediovestibular ankylosis
* radiological confirmation if CT-scan before inclusion available

Exclusion Criteria:

* Individuals not covered by the french public health insurance
* Pure-tone average < 30 dB ou > 90 dB
* Programmed stapes surgery during the observation period
* Previous treatment by biphosphonate
* Known intolerance to tiludronate
* Other contraindications to tiludronate treatment:
* allergy to biphosphonates
* hypersensitivity to one of the excipients
* severe renal failure (creatinine clearance < 30 mL/min)
* juvenile Paget's disease
* pregnancy and breastfeeding
* galactose intolerance, lactase insufficiency, glucose-galactose malabsorption
* Ongoing chemotherapy or radiotherapy or patient achieves of a cancer
* Long-term systemic steroid treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Hearing preservation on pure-tone audiometry at 2 years | year 2
  Effect on hearing preservation as assessed by air conduction pure-tone average at 2 years.
  Hearing deterioration is defined by a deterioration of pure-tone average by air conduction >20 dB at 500, 1000, 2000 and 4000 Hz between inclusion and the end of the observation period.

SECONDARY OUTCOMES:
hearing preservation at one year | year 1
  Effect on hearing preservation as assessed by air conduction pure-tone average at 1 year
cochlear function | years 1 and 2
  Effect on cochlear function preservation as evaluated by bone conduction pure-tone average (500, 1000, 2000 and 4000 Hz) at 1 and 2 years.
Stapedial reflex preservation | years 1 and 2
  Percentage of stapedial reflex preservation on the controlateral ear if unilateral otosclerosis at 1 and 2 years.
Speech reception threshold and speech discrimination score | years 1 and 2
  Effect on speech reception threshold ans speech discrimination score at 1 and 2 years.
Tinnitus and balance disorders | years 1 and 2
  Effect on the prevalence and the intensity of tinnitus and balance disorders as evaluated by questionnary at 1 and 2 years.
Radiological bone density | year 2
  Effect on radiological bone density at fissula ante fenestram as assessed on high resolution temporal bone CT-scans before and after treatment by calculation of fissula ante fenestram / temporal bone squama cortex bone density ration on axial views.
Tolerance | month 3
  Clinical tolerance during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexis BOZORG-GRAYELI, Pr, Principal Investigator — Hôpital Général, CHU de Dijon
Locations (1):
- Beaujon Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No